CLINICAL TRIAL: NCT04529356
Title: A Randomized Controlled Study of Transcranial Magnetic Stimulation for Postoperative Headache in Patients With Growth Hormone（GH） Pituitary Tumor
Brief Title: The TMS Treatment for Postoperative Headache in GH Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2020-844
Record Dates: First submitted 2020-08-07; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Headache; Pituitary Tumor; Acromegaly
MeSH Terms: conditions — Headache; Pituitary Neoplasms; Acromegaly | interventions — Transcranial Magnetic Stimulation; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simple acetaminophen treatment (Sham Comparator): Acetaminophen will be taken when patients suffered from headache during the study. No specific dosage and frequency was required for this group as long as the participants record the exact drug usage.
  Interventions: Drug: Acetaminophen
- Simple acetaminophen combined with low-frequency rTMS (Active Comparator): Apart from acetaminophen usage, low frequency TMS (1HZ) will be used in patients three times a month for 6 months.
  Interventions: Device: Transcranial magnetic stimulation; Drug: Acetaminophen
- Simple acetaminophen combined with high-frequency rTMS (Experimental): Apart from acetaminophen usage, high frequency TMS (10HZ) will be used in patients three times a month for 6 months.
  Interventions: Device: Transcranial magnetic stimulation; Drug: Acetaminophen

INTERVENTIONS:
Device: Transcranial magnetic stimulation — By using different frequency of TMS, the device can generate different effects. For low frequency, such as 1HZ, it mainly generates inhibition on the brain cortex; while high frequency (usually higher than 10HZ) can generate stimulation effects. The later one could be used to treat different central nervous disease.
  Arms: Simple acetaminophen combined with high-frequency rTMS; Simple acetaminophen combined with low-frequency rTMS
Drug: Acetaminophen — Acetaminophen is used as the painkiller to alleviate patients' headache before and during the clinical trial. In order to decrease the medication bias, we required these patients to only use acetaminophen instead of other non-steroid anti-inflammatory drugs. In the meantime, participants are requested to recorder the frequency and dosage of acetaminophen they used during the treatment course.

SUMMARY:
Headache is a very common main complaint of patients with GH pituitary tumor, which has seriously affected the normal work and life of patients. Although the current surgery and drugs have a certain effect on patients with headache, the overall effect is not satisfied. However, the use of COX-2 inhibitors, non-steroidal anti-inflammatory drugs and other analgesics are only effective for some patients with headaches, and long-term use has adverse reactions. Therefore, it is necessary to seek new treatments for postoperative headaches in patients with GH pituitary tumors. Transcranial magnetic stimulation (TMS) modulates the excitability of the underlying cerebral cortex by applying a rapidly changing magnetic field on the surface of the scalp. It is a relatively simple and safe method. It is currently approved for treating depression, migraine, obsessive-compulsive disorder, and Alzheimer's disease. Several small clinical studies have proven that rTMS can be used to prevent and treat Headache. Therefore, this study aims to observe the efficacy and safety of TMS in the treatment of postoperative headache in patients with GH pituitary tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GH tumor who have undergone transnasal pituitary tumor resection or craniotomy for pituitary tumor resection in the past (3 months or more), aged between 18 and 60 years old, regardless of gender;

  * Preoperative glucose tolerance test (OGTT) simultaneously determines that the trough value of GH is greater than 1ng/ml, and the level of IGF-1 is greater than the upper limit of the age-sex-matched normal value; ③. Biochemical remission is achieved after surgery, that is, the random GH value is less than 1ng/ml, and the IGF-1 level is within the normal range of age and gender matching; ④. The patient still has headaches after the operation, the duration of each attack is more than 4 hours, and the attack is more than 3 times per month; ⑤. The patient is in a headache attack period; ⑥. A clear consciousness, able to understand and sign an informed consent form.

Exclusion Criteria:

* Patients who are being treated with somatostatin and bromocriptine;

  * Patients with other intracranial organic diseases;

    * Pregnant women and children who cannot express;

      * Patients with other malignant tumors;

        * Participate in other clinical research in the same period; ⑥. Patients with severe medical complications, such as heart, lung, kidney, liver and other diseases, severe hypertension or poor blood pressure control, hyperglycemia, blood diseases;

          * Those with mental illness who cannot cooperate well with the experiment;

            * Patients with acute infection or open wounds; ⑨. Acetaminophen is contraindicated (hemolytic anemia, severe liver and kidney dysfunction) or allergic to its components; ⑩. Patients with contraindications to transcranial magnetic stimulation: patients or users who have implanted cardiac pacemakers, implantable defibrillators and neurostimulators together; those who have a history of epilepsy; wear electronic products (such as insulin Pumps, Holter, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
changes in the degree of headache | 6 months
  The degree of headache will be measured by the Visual Analog Scale VAS and the scores change before and after 6 months of intervention will be compared among 3 groups
the improvement of quality of life(QOL) | 6 months
  Migraine Defect Assessment Questionnaire MIDAS will be used to evaluate QOL. The QOL will be assessed before and after 6 months of intervention and the changes of MIDAS scores will be compared among 3 groups

SECONDARY OUTCOMES:
The decrease of using acetaminophen | 6 months
  During the experiment, patients will be required to record the dosage of acetaminophen they used. Our anticipated secondary outcome is the decreased usage of painkiller in the rTMS treated patients.The total dosage of acetaminophen used in 1st month and the 6th month during the study will be recorded and the changes of the dosage will be compared among the 3 groups.